CLINICAL TRIAL: NCT07310615
Title: Mindfulness-Based Psychoeducation Improves Mindfulness and Medication Adherence in Schizophrenia: A Randomized Controlled Trial
Brief Title: Mindfulness Psychoeducation for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer USLU (Other)
Responsible Party: Sponsor-Investigator, Ömer USLU, Dr. Ömer Uslu, PhD - Principal Investigator, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMER-RCT-2025-SCH
Record Dates: First submitted 2025-12-09; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mindfulness; Psychoeducation; Randomized Controlled Trial
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the experimental group (mindfulness-based psychoeducation) or the control group with no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Psychoeducation (Experimental): Participants will receive an 8-session mindfulness-based psychoeducation program.
  Interventions: Behavioral: Mindfulness-Based Psychoeducation Program
- Control: Routine Care (Active Comparator): Participants in this arm will receive Routine Care provided by the psychiatric outpatient clinic. Routine Care includes standard follow-up, medication management, and usual clinical monitoring. No additional psychoeducation or mindfulness-based intervention will be provided during the study period.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: Mindfulness-Based Psychoeducation Program — A structured 8-session mindfulness-based psychoeducation program including mindfulness exercises, psychoeducation, breathing techniques and adherence-support strategies.
  Arms: Mindfulness-Based Psychoeducation
Other: Routine Care — Standard outpatient psychiatric care delivered by the clinic. No additional psychoeducation or mindfulness intervention is provided.
  Arms: Control: Routine Care

SUMMARY:
This study aims to examine the effects of a mindfulness-based psychoeducation program on mindfulness levels and treatment adherence among individuals diagnosed with schizophrenia. Schizophrenia is a chronic psychiatric disorder that affects thinking, emotions, and behavior, and difficulties in adhering to prescribed treatments are commonly observed. Poor treatment adherence is associated with relapse, increased hospitalization, and reduced overall functioning.

This randomized controlled study includes 40 patients assigned to either an experimental group or a control group. The experimental group receives a structured mindfulness-based psychoeducation program, while the control group receives treatment as usual without any additional intervention. Assessments are conducted before and after the intervention using a Personal Information Form, a Mindfulness Scale, and the Morisky Medication Adherence Scale.

DETAILED DESCRIPTION:
Schizophrenia is a severe and chronic psychiatric disorder characterized by disturbances in thought processes, perceptions, emotions, and behaviors. Despite advances in pharmacological and psychosocial treatments, maintaining long-term treatment adherence remains a major challenge in the management of schizophrenia. Non-adherence to treatment is associated with adverse clinical outcomes, including relapse, rehospitalization, impaired functioning, and increased healthcare utilization.

Mindfulness-based interventions have been increasingly applied in mental health settings to support awareness of internal experiences, emotional regulation, and stress management. Mindfulness practices may contribute to treatment engagement by enhancing individuals' awareness of symptoms, daily routines, and coping responses. Psychoeducation is a core component of psychiatric nursing care and focuses on improving knowledge about illness, treatment processes, and coping strategies. Integrating mindfulness practices into a psychoeducation framework may offer a structured approach to supporting treatment engagement in individuals with schizophrenia.

Study Purpose

The primary purpose of this randomized controlled trial is to evaluate the effects of a structured mindfulness-based psychoeducation program on:

Mindfulness levels Treatment adherence among individuals diagnosed with schizophrenia. Study Design

This study uses a randomized controlled experimental design with pre-test and post-test measurements. Participants are randomly assigned to one of two groups:

Experimental group: Receives a structured mindfulness-based psychoeducation program delivered in weekly sessions.

Control group: Receives treatment as usual without additional intervention during the study period.

The intervention is designed to be applicable within routine psychiatric care settings and includes structured content focusing on mindfulness awareness, psychoeducation related to illness and treatment, and skill development.

Participants A total of 40 individuals diagnosed with schizophrenia are included in the study, with 20 participants in the experimental group and 20 in the control group. Participants are recruited from psychiatric outpatient clinics. Inclusion criteria include a clinical diagnosis of schizophrenia, clinical stability as determined by the treating psychiatrist, and sufficient cognitive capacity to participate in the intervention. Exclusion criteria include active psychotic symptoms, acute hospitalization, severe neurological disorders, or inability to provide informed consent.

Intervention Description

The mindfulness-based psychoeducation program consists of structured sessions delivered over a defined period. Each session includes:

Introduction to mindfulness concepts Guided mindfulness practices (e.g., breathing awareness, body scan, grounding exercises) Psychoeducation related to illness understanding, symptom management, and treatment processes Group discussion and reflection activities Homework assignments to support daily mindfulness practice The program is structured to support awareness of internal experiences, recognition of symptoms, and engagement with treatment routines.

Outcome Measures

Data are collected using the following instruments:

Mindfulness Scale: To assess levels of mindful awareness Morisky Medication Adherence Scale: To assess treatment adherence Personal Information Form: To collect demographic and clinical characteristics Measurements are obtained at baseline (pre-test) and after completion of the intervention (post-test).

Data Analysis Quantitative data analyses include descriptive statistics and comparisons of pre-test and post-test scores within and between groups using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-5 criteria
* Age between 18-65 years
* Being clinically stable for at least the past 3 months
* Able to communicate, read, and understand Turkish
* Receiving outpatient psychiatric follow-up
* Willingness to participate and providing informed consent

Exclusion Criteria:

* Presence of acute psychotic symptoms requiring immediate hospitalization
* Comorbid intellectual disability, neurological disorder, or severe cognitive impairment
* Substance or alcohol dependence within the last 6 months
* Participation in any mindfulness-based or psychoeducational program within the last year
* Severe visual or hearing impairment preventing participation
* Any condition judged by the clinician to contraindicate participation in group sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
Mindfulness level (Mindful Attention Awareness Scale) | Baseline and 8 weeks after intervention
  Mindfulness was assessed using the Mindful Attention Awareness Scale (MAAS). Score range: 15-90. Higher scores indicate greater mindfulness.

SECONDARY OUTCOMES:
Mindfulness level at 8 weeks (Mindful Attention Awareness Scale) | 8 weeks
  Description:
  Mindfulness was assessed using the Mindful Attention Awareness Scale (MAAS). Score range: 15-90. Higher scores indicate greater mindfulness.
Self-compassion level at 8 weeks (Self-Compassion Scale) | 8 weeks
  Self-compassion was assessed using the Self-Compassion Scale (SCS). Score range: 26-130. Higher scores indicate greater self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Uslu, PhD, RN, Principal Investigator — Söke Fehime Faik Kocagöz Hospital
Locations (1):
- Söke Fehime Faik Kocagöz State Hospital, Aydin, Söke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to ethical and institutional restrictions. The dataset includes sensitive health information from patients diagnosed with schizophrenia, and the informed consent process did not include permission for public data sharing. Therefore, in accordance with privacy regulations and ethical committee requirements, IPD will not be made available to other researchers